CLINICAL TRIAL: NCT03538860
Title: A Clinical Trial to Validate an Automated Online Language Interpreting Tool With Hispanic Patients Who Have Limited English Proficiency - Phase Two.
Brief Title: Validation of an Automated Online Language Interpreting Tool - Phase Two.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1131922; R01HS024949 (AHRQ)
Record Dates: First submitted 2018-03-01; First posted 2018-05-29 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Mood Disorder; Anxiety Disorder; Substance Use Disorder; Chronic Medical Condition
Keywords: Telepsychiatry; AsynchronousTelepsychiatry; Automated Translation
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Method A first then Method B (Other): Conventional in-person interview with a psychiatrist with a live human interpreter with crossover to asynchronous telepsychiatry
  Interventions: Behavioral: Active comparator: Human interpreter; Behavioral: Intervention: Asynchronous Telepsychiatry
- Method B first then Method A (Other): Asynchronous telepsychiatry - that is, video-recorded interviews that are subsequently processed with automated speech recognition and machine translation technologies, with crossover to conventional in-person interview with a psychiatrist with a live human interpreter
  Interventions: Behavioral: Active comparator: Human interpreter; Behavioral: Intervention: Asynchronous Telepsychiatry

INTERVENTIONS:
Behavioral: Active comparator: Human interpreter — A Spanish-speaking patient is diagnostically assessed in-person by an English-speaking psychiatrist through a Spanish-speaking interpreter.
Behavioral: Intervention: Asynchronous Telepsychiatry — A Spanish-speaking patient is interviewed in Spanish by a trained mental health interviewer. The interview is video-recorded in real-time, automatically translated into English with sub-titles added to the video file, and sent to a psychiatrist and to 3 English-speaking psychiatrists to asynchronously review the video and make a diagnosis.

SUMMARY:
There is a pressing national need to provide higher-quality, more effectively accessible language interpretation services to improve the health outcomes of Americans who have limited English proficiency (LEP). This project addresses a critical component of this problem: The need to improve access to high quality, mental health services for diverse populations by improving the flow of clinical work across care settings (primary care and specialty care) through the use of innovative online asynchronous methods of language interpretation and clinical communication. The investigators are conducting a two phase study. The first phase is completed and involved developing and testing the interpreting tool. The second phase of the research is a clinical trial to compare two methods of cross-language psychiatric assessment.

DETAILED DESCRIPTION:
The investigators propose to develop and test a novel automated asynchronous interpretation tool. The proposed project builds on previous research, piloting the automated asynchronous interpretation tool. This 5-year project will be conducted in two phases. In Phase 1 the investigators iteratively evaluate and refine the automated asynchronous interpretation tool already developed in prior studies. In Phase 2, the investigators evaluate this tool using a two-group randomized cross-over trial. Investigators compare:

* Method A (current gold standard of in-person real-time interpreting practice). A Spanish-speaking patient is diagnostically assessed in-person by an English-speaking psychiatrist through a Spanish-speaking interpreter.
* Method B (comparative practice - ATP). A Spanish-speaking patient is interviewed in Spanish by a trained mental health interviewer. The interview is recorded in real time, translated into English using the automatic interpretation tool and adding sub-titles to the video file, and sent to an English-speaking psychiatrist to asynchronously - that is, at a later time - review the video and make a diagnosis.

All patients will undergo evaluation by both methods. Half of the patients will be randomized to be assessed by Method A first, followed by Method B and half to be assessed by Method B first, followed by Method A. The specific aims of the study are :

* Aim 1: To iteratively evaluate and refine the automated asynchronous interpretation tool already developed in prior studies.
* Aim 2: To compare patient satisfaction of Method A vs. Method B.
* Aim 3: To compare the diagnostic accuracy and psychiatrist inter-rater reliability of Method A vs. Method B and demonstrate psychiatrist inter-rater reliability for Method B.
* Aim 4: To compare the interview and language interpretation quality and accuracy of Method A vs. Method B.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria: Hispanic patients with significant Limited English proficiency (LEP)

* aged 18 or older
* diagnosis of a mood disorder, anxiety disorder, or substance/alcohol abuse disorder(s)
* Diagnosis of a chronic medical condition
* referred by PCP or self-referral with PCP informed

Exclusion Criteria: Criteria:

* less than 18 years
* imminent suicidal ideation and/or plans
* immediate violent intentions or plans
* significant cognitive deficits
* patient who's PCP recommends not participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Measured at one time point by each psychiatrist, once both methods of interviews are completed in one day
  Diagnosis accuracy with respect to gold standard SCID for Method B will be evaluated against Method A.
Diagnostic Inter-rater reliability | Measured at one time point by each psychiatrist, once both methods of interviews are completed in one day
  Using independent assessments from four psychiatrists for each of the 100 method B interviews the investigators will also examine inter-rater reliability of Method B diagnosis.

SECONDARY OUTCOMES:
Satisfaction ratings | Measured at one time point by each psychiatrist, once both methods of interviews are completed in one day
  Satisfaction ratings from patients' questionnaires
Interview and language interpretation quality | Measured at one time point by each psychiatrist, once both methods of interviews are completed in one day
  All 200 interviews in both methods will be video recorded and the audio transcribed. The investigators will measure and compare the two interview methods interpretation quality through perception of interpretation quality
Interview and language interpretation accuracy | Measured at one time point by each psychiatrist, once both methods of interviews are completed in one day
  All 200 interviews in both methods will be video recorded and the audio transcribed. The investigators will measure and compare the two interview methods accuracy through the presence of medical errors, and the presence of language errors

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tougas H, Chan S, Shahrvini T, Gonzalez A, Chun Reyes R, Burke Parish M, Yellowlees P. The Use of Automated Machine Translation to Translate Figurative Language in a Clinical Setting: Analysis of a Convenience Sample of Patients Drawn From a Randomized Controlled Trial. JMIR Ment Health. 2022 Sep 6;9(9):e39556. doi: 10.2196/39556. PMID 36066959
- [Derived] Parish MB, Gonzalez A, Hilty D, Chan S, Xiong G, Scher L, Liu D, Sciolla A, Shore J, McCarron R, Kahn D, Iosif AM, Yellowlees P. Asynchronous Telepsychiatry Interviewer Training Recommendations: A Model for Interdisciplinary, Integrated Behavioral Health Care. Telemed J E Health. 2021 Sep;27(9):982-988. doi: 10.1089/tmj.2020.0076. Epub 2021 Jan 12. PMID 33434453

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03538860/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03538860/ICF_001.pdf